CLINICAL TRIAL: NCT03777033
Title: Systematic Administration vs on Demand Administration of Calcium and Vitamin D After Thyroidectomy. A Randomized Control Trial
Brief Title: Systematic Administration of Calcium and Vitamin D After Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hellenic Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Sophocles Lanitis, M.D, PhD, Consultant in General Surgery, Hellenic Red Cross Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ca/vitD in thyroidectomy
Record Dates: First submitted 2017-10-25; First posted 2018-12-17 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Diseases
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Intervention Model Description: Randomized control trial - control group ( supplements of calcium and vit D on demand) vs study group ( systematic administration of oral calcium and vit D )
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Patients after thyroidectomy will be managed as usual. Oral or IV supplements of Calcium will be giver on demand and recorded according to the clinical picture or the biochemical hypocalcaemia.
- Study group (Experimental): Intervention: the patients will be given prophylactically ca and vit D. Patients after thyroidectomy will be given systematically from the day of operation a scheme with oral calcium in the form of 1000ca++mg/tab and oral alfacalcidol in the form of 0.5 micrograms/tb Intervention: The patients will receive one tablet three times a day oral calcium (3g/d) and 2 tablets , two times a day alfacalcidiol (2 micrograms/d) for the first 5 days. Afterwards they will be taking 2 tablets a day of oral calcium ( 2g) and 2 tablets a day alfacalcidiol (1micrograms/d) for another 10 days ( total 15 days)
  Interventions: Drug: Prophylactic protocol with Ca and Vit D

INTERVENTIONS:
Drug: Prophylactic protocol with Ca and Vit D — 3g calcium /day for 5 days and then 2g/day for 10 days 2 Micrograms Alfacalcidol/day and then 1 microgram /day for 10 days
  the Prophylactic protocol with Ca and Vit D will be given in the form of Alfacalcidol 0.5 Micrograms Capsule and CALCIUM CARBONATE + CALCIUM GALACTOGLUCONATE 1000mg tablet
  Other Names: one-alfa and mega calcium
  Arms: Study group

SUMMARY:
Transient hypocalcaemia consist the most common postoperative complication after thyroidectomy (10-45%). It may be mild and subclinical or cause mild or severe symptoms and may lead to longer hospital stay as well as in discomfort of the patients. For the management oral or intravenous calcium with or without vitamin D administration can be used based on the blood calcium levels and on the symptomatology. The investigators intent to study a new protocol with oral calcium and vitamin D given systematically from the day of operation to assess if this practice can minimize the rate of transient hypocalcaemia and as a consequence minimize the length of stay in the hospital.

DETAILED DESCRIPTION:
Transient hypocalcaemia consist the most common postoperative complication after thyroidectomy (10-45%). It may be mild and subclinical or cause mild or severe symptoms and may lead to longer hospital stay as well as in discomfort of the patients. For the management oral or intravenous calcium with or without vitamin D administration can be used based on the blood calcium levels and on the symptomatology.

Group A = control group will be managed as usual. Oral or IV supplements of Calcium will be giver on demand and recorded according to the clinical picture or the biochemical hypocalcaemia.

Group B= study group will be given systematically from the day of operation a scheme with oral calcium in the form of 1000ca++mg/tab and oral alfacalcidol in the form of 0.5 micrograms/tb The patients will receive one tablet three times a day oral calcium (3g/d) and 2 tablets , two times a day alfacalcidiol (2 micrograms/d) for the first 5 days. Afterwards they will be taking 2 tablets a day of oral calcium ( 2g) and 2 tablets a day alfacalcidiol (1micrograms/d) for another 10 days ( total 15 days) The investigators intent to minimize the immediate transient hypocalcaemia rate and give time to the parathyroids which may have been bruised or have compromised function initially to recover by day 15.

The 1st and 2nd postoperative day the invastigators are going to take blood samples and assess the 25 hydroxy vit D, the parathyroid hormone (PTH) and the Ca++. The investigators will also assess the calcium levels after the first week and if necessary ( in cases with longstanding hypocalcaemia ) in later day.

The patients will be discharged from the hospital the day after the operation provided the calcium levels are within normal range and they are completely asymptomatic.

In case of symptoms after the discharge the patients will be managed accordingly and this will be recorded in the records of each patient

ELIGIBILITY:
Inclusion Criteria:

* Thyroid pathology only
* No calcium metabolism problems
* Total / near total thyroidectomy

Exclusion Criteria:

* Renal failure,
* Secondary hyperparathyroidism,
* Primary hyperparathyroidism,
* thyroid lobectomy,
* Thyroid reoperation

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-03-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-08-04 (Estimated)

PRIMARY OUTCOMES:
blood calcium levels (mg/dl) on the 1st postoperative day | From the end of the operation until 24 hours after the operation
  blood calcium measured in a blood sample in mg/dl
blood calcium levels (mg/dl) on the 2nd postoperative day | From the end of the operation until 48 hours after the operation
  blood calcium measured in a blood sample in mg/dl
Length of hospital stay in days | From the day of the operation until a week after the operation
  how many days the patient remained in the hospital

SECONDARY OUTCOMES:
Overall cost of the treatment ( euros) | From the day of the operation until a month from the operation
  how did this practice affected the cost of treatment of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Sophocles Lanitis, Principal Investigator — Korgiallenio benakeio hellenic red cross hospital
Locations (1):
- "Korgialenio-Benakio", Hellenic Red Cross Athens General Hospital,, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Effectiveness of preventative and other surgical measures on hypocalcemia following bilateral thyroid surgery: a systematic review and meta-analysis. — https://www.ncbi.nlm.nih.gov/pubmed/25203484
- See also: Role of postoperative vitamin D and/or calcium routine supplementation in preventing hypocalcemia after thyroidectomy: a systematic review and meta-analysis. — https://www.ncbi.nlm.nih.gov/pubmed/23635556